CLINICAL TRIAL: NCT03017716
Title: Inflammatory Back Pain and Gluten Free Diet
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, MD, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACPM14
Record Dates: First submitted 2016-12-30; First posted 2017-01-11 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Back Pain
Keywords: Inflammatory back pain; gluten-free diet; celiac disease; non-celiac wheat sensitivity
MeSH Terms: conditions — Celiac Disease | interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBP patients on standard therapy (No Intervention): IBP patients on standard therapy.
- IBP patients on standard therapy and GFD (Active Comparator): IBP patients on standard therapy and GFD
  Interventions: Other: Gluten free diet

INTERVENTIONS:
Other: Gluten free diet — The investigators will evaluate the effect of a gluten free diet (GFD) in IBP patients, randomly assigned to receive standard therapy for IBP or standard therapy for IBP plus GFD, for a period of at least one year.
  Arms: IBP patients on standard therapy and GFD

SUMMARY:
Articular involvement is the most frequent extra-intestinal manifestation of inflammatory bowel diseases (IBD). IBD-related spondyloarthropathy is mainly characterised by axial involvement (including inflammatory back pain, isolated sacroiliitis and ankylosing spondylitis) but may also be associated with peripheral symptoms (i.e peripheral arthritis, dactylitis and enthesopathy, such as Achilles tendinitis, plantar fasciitis, and chest wall pain). In particular, inflammatory back pain (IBP) is characterised by an insidious onset, improves after exercise but not with rest, and is associated with morning stiffness. Up to now, several criteria sets have been proposed to define IBP. Studies conducted in various populations have confirmed a high sensitivity and specificity for the Berlin criteria. Celiac disease (CD) is an autoimmune systemic disease having among its clinical manifestations frequent symptoms common to rheumatologic diseases. Recently, it has been reported that a consistent percentage of the general population consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have CD or wheat allergy. This clinical condition has been named Non-Celiac Gluten Sensitivity' (NCGS) or Non-celic Wheat Sensitivity (NCWS). The clinical picture of NCWS is characterized by combined gastrointestinal and extra-intestinal or systemic manifestations. Many patients affected with CD and NCWS complain of IBP-like symptoms, which generally improve, together with the other clinical manifestations of the diseases, during a gluten-free diet (GFD). Therefore, the aims of the present study are to investigate 1) the effect of a GFD in IBP patients, randomly assigned to receive standard therapy for IBP or standard therapy for IBP plus GFD, for a period of at least one year, and 2) the prevalence of IBP in CD and in NCWS patients.

DETAILED DESCRIPTION:
Articular involvement is the most frequent extra-intestinal manifestation of inflammatory bowel diseases (IBD), frequently follows a course that is independent of the course of intestinal involvement, and its diagnosis mainly relies on clinical evidence and imaging data, because laboratory assessments are rarely useful. More in details, IBD-related arthropathy is one of a group of inflammatory arthritides, known as seronegative spondyloarthropathies, that also includes idiopathic ankylosing spondylitis, reactive arthritis, psoriatic arthritis, and undifferentiated seronegative spondyloarthropathies, all of which are classified on the basis of peripheral arthritis (asymmetrical, predominantly in the lower extremities) and/or inflammatory spinal involvement in IBD patients using the well-known criteria of the European Spondyloarthropathy Study Group. IBD-related spondyloarthropathy is mainly characterised by axial involvement (including inflammatory back pain, isolated sacroiliitis and ankylosing spondylitis) but may also be associated with peripheral symptoms (i.e peripheral arthritis, dactylitis and enthesopathy, such as Achilles tendinitis, plantar fasciitis, and chest wall pain). In particular, inflammatory back pain (IBP) is characterised by an insidious onset, improves after exercise but not with rest, and is associated with morning stiffness. It may also present as pain during the second half of the night and/or alternating buttock pain. Up to now, several criteria sets have been proposed to define IBP. Firstly, the Calin criteria set was developed in 1977 and has since then been most widely used for defining IBP. The Calin criteria set has no entry criteria and is not based on standardized questions. Studies conducted in various populations have confirmed a high sensitivity for the Calin criteria, but shown much lower specificity than that reported in the original study. Berlin criteria for IBP were derived from a controlled study, including patients with ankylosing spondylitis and mechanical low back pain, who all had chronic low back pain. Berlin criteria are applicable only to those patients with chronic low back pain (>3 months) and age younger than <50 years old. This criteria set yielded a sensitivity of 70% and a specificity of 81% if at least two of the four following criteria were met: morning stiffness of >30-min duration, improvement in back pain with exercise but not with rest, awakening because of back pain during the second half of the night only, and alternating buttock pain. Assessment of Spondyloarthritis International Society (ASAS) has just recently published new criteria for classification of IBP. These were based on the expert judgment of the rheumatologist as the "gold standard" for diagnosing IBP in patients with chronic back pain of unknown origin. These new candidate IBP criteria administered by the interviewing clinician included the domains "improvement with exercise," "nocturnal pain," "age at onset <40 years," and "no improvement with rest." They were then validated in a distinct cohort of patients presenting to the rheumatologist with new-onset back pain and were shown to have a sensitivity of 79.6% and specificity of 72.4%. Celiac disease (CD) is an autoimmune systemic disease having among its clinical manifestations frequent symptoms common to rheumatologic diseases, such as musculoskeletal pain, asthenia, and cognitive fatigue. Recently, it has been reported that a consistent percentage of the general population consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have CD or wheat allergy. This clinical condition has been named Non-Celiac Gluten Sensitivity' (NCGS). In a previous paper the investigators suggested the term 'Non-Celiac Wheat Sensitivity' (NCWS), since it is not known what component of wheat causes the symptoms in NCGS patients, and the investigators also showed that these patients had a high frequency of coexistent multiple food hypersensitivity. The clinical picture of NCWS is characterized by combined gastrointestinal (bloating, abdominal pain, diarrhea and/or constipation, nausea, epigastric pain, gastroesophageal reflux, aphthous stomatitis) and extra-intestinal or systemic manifestations (headache, depression, anxiety, 'foggy mind,' tiredness, dermatitis or skin rash, fibromyalgia-like joint/muscle pain, leg or arm numbness, and anemia). NCWS lacks of specific diagnostic tests, being its diagnosis essentially of exclusion. Many patients affected with CD and NCWS complain of IBP-like symptoms, which significantly affect the patients' quality of life and generally improve, together with the other clinical manifestations of the diseases, during a gluten-free diet (GFD). Therefore, the aims of the present study are to investigate 1) the effect of a GFD in IBP patients, randomly assigned to receive standard therapy for IBP or standard therapy for IBP plus GFD, for a period of at least one year, and 2) the prevalence of IBP in CD and in NCWS patients.

ELIGIBILITY:
Inclusion Criteria:

To diagnose IBP the standard Berlin Criteria will be adopted. IBP is defined by at least 2 positive responses among four items:

* morning stiffness >30 min of duration
* improvement in back pain with exercise but not with rest
* awakening because of back pain during the second half of the night only
* alternating buttock pain.

To diagnose CD the standard criteria will be adopted. All the patients will meet the following criteria:

* positive serum anti-transglutaminase (anti-tTG) and anti-endomysium (EmA) immunoglobulin (Ig)A and IgG antibodies
* presence of intestinal villous atrophy.

To diagnose NCWS the recently proposed criteria will be adopted. All the patients will meet the following criteria:

* negative serum anti-transglutaminase (anti-tTG) and anti-endomysium (EmA) immunoglobulin (Ig)A and IgG antibodies
* absence of intestinal villous atrophy
* negative IgE-mediated immune-allergy tests to wheat (skin prick tests and/or serum specific IgE detection)
* resolution of the IBS symptoms on standard elimination diet, excluding wheat, cow's milk, egg, tomato, chocolate, and other self-reported food(s) causing symptoms
* symptom reappearance on double-blind placebo-controlled (DBPC) wheat challenge. As the investigators previously described in other studies, DBPC cow's milk protein challenge and other "open" food challenges will be performed too.

Exclusion Criteria:

Exclusion criteria for NCWS diagnosis will be:

* positive EmA in the culture medium of the duodenal biopsies, also in the case of normal villi/crypts ratio in the duodenal mucosa
* self-exclusion of wheat from the diet and refusal to reintroduce it before entering the study
* other previously diagnosed gastrointestinal disorders
* other previously diagnosed rheumatic diseases
* nervous system disease and/or major psychiatric disorder
* physical impairment limiting physical activity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal (back pain) evaluation at baseline and after GFD | Change from baseline at 12 months
  Musculoskeletal (back pain) evaluation, from baseline at 12 months of GFD, according to the scores calculated on the basis of Visual Analogue Scales for Musculoskeletal (back pain), taking into account whether the patients adhered or not to the GFD.
Changes in cytokines production from peripheral blood mononuclear (PBMC) at baseline and after GFD | Change from baseline at 12 months
  Changes in cytokines production from peripheral blood mononuclear (PBMC), from baseline (i.e. at diagnosis) at 12 months of GFD, taking into account whether the patients adhered or not to the GFD.

SECONDARY OUTCOMES:
Prevalence of IBP in CD and in NCWS patients. | up to 12 months
  Prevalence of IBP in CD and in NCWS patients.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, PhD, Study Director — University of Palermo
Locations (2):
- Italy (2):
  - Department of Internal Medicine, Giovanni Paolo II Hospital of Sciacca, Sciacca, Agrigento
  - Department of Internal Medicine, University Hospital of Palermo, Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Role of FODMAPs in Patients With Irritable Bowel Syndrome. Nutr Clin Pract. 2015 Oct;30(5):665-82. doi: 10.1177/0884533615569886. Epub 2015 Feb 18. PMID 25694210
- [Result] Carroccio A, D'Alcamo A, Mansueto P. Nonceliac wheat sensitivity in the context of multiple food hypersensitivity: new data from confocal endomicroscopy. Gastroenterology. 2015 Mar;148(3):666-7. doi: 10.1053/j.gastro.2014.11.047. Epub 2015 Jan 24. No abstract available. PMID 25625764
- [Result] Carroccio A, Soresi M, D'Alcamo A, Sciume C, Iacono G, Geraci G, Brusca I, Seidita A, Adragna F, Carta M, Mansueto P. Risk of low bone mineral density and low body mass index in patients with non-celiac wheat-sensitivity: a prospective observation study. BMC Med. 2014 Nov 28;12:230. doi: 10.1186/s12916-014-0230-2. PMID 25430806
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Non-celiac gluten sensitivity: literature review. J Am Coll Nutr. 2014;33(1):39-54. doi: 10.1080/07315724.2014.869996. PMID 24533607
- [Result] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Result] Carroccio A, Mansueto P, D'Alcamo A, Iacono G. Non-celiac wheat sensitivity as an allergic condition: personal experience and narrative review. Am J Gastroenterol. 2013 Dec;108(12):1845-52; quiz 1853. doi: 10.1038/ajg.2013.353. Epub 2013 Nov 5. PMID 24169272
- [Result] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Result] Carroccio A, Brusca I, Mansueto P, D'alcamo A, Barrale M, Soresi M, Seidita A, La Chiusa SM, Iacono G, Sprini D. A comparison between two different in vitro basophil activation tests for gluten- and cow's milk protein sensitivity in irritable bowel syndrome (IBS)-like patients. Clin Chem Lab Med. 2013 Jun;51(6):1257-63. doi: 10.1515/cclm-2012-0609. PMID 23183757
- [Result] Dougados M, van der Linden S, Juhlin R, Huitfeldt B, Amor B, Calin A, Cats A, Dijkmans B, Olivieri I, Pasero G, et al. The European Spondylarthropathy Study Group preliminary criteria for the classification of spondylarthropathy. Arthritis Rheum. 1991 Oct;34(10):1218-27. doi: 10.1002/art.1780341003. PMID 1930310
- [Result] Calin A, Porta J, Fries JF, Schurman DJ. Clinical history as a screening test for ankylosing spondylitis. JAMA. 1977 Jun 13;237(24):2613-4. PMID 140252
- [Result] Rudwaleit M, Metter A, Listing J, Sieper J, Braun J. Inflammatory back pain in ankylosing spondylitis: a reassessment of the clinical history for application as classification and diagnostic criteria. Arthritis Rheum. 2006 Feb;54(2):569-78. doi: 10.1002/art.21619. PMID 16447233
- [Result] Sieper J, van der Heijde D, Landewe R, Brandt J, Burgos-Vagas R, Collantes-Estevez E, Dijkmans B, Dougados M, Khan MA, Leirisalo-Repo M, van der Linden S, Maksymowych WP, Mielants H, Olivieri I, Rudwaleit M. New criteria for inflammatory back pain in patients with chronic back pain: a real patient exercise by experts from the Assessment of SpondyloArthritis international Society (ASAS). Ann Rheum Dis. 2009 Jun;68(6):784-8. doi: 10.1136/ard.2008.101501. Epub 2009 Jan 15. PMID 19147614